CLINICAL TRIAL: NCT05792670
Title: Can High Ventilation Mode Achieve Higher Success Rates in Retrograde Intrarenal Surgery? Single-Blind Randomized, Prospective, Single-Center Study
Brief Title: Can High Ventilation Provide Higher Success Rates in Retrograde Intrarenal Surgery?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Namik Kemal University (Other)
Responsible Party: Principal Investigator, Cagri DOGAN, Assistant.Prof, Namik Kemal University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 2022.179.10.03
Record Dates: First submitted 2023-03-01; First posted 2023-03-31 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Kidney; Mobile
Keywords: renal mobility; urinary stone; mechanic ventilation; success status
MeSH Terms: conditions — Urinary Calculi

STUDY DESIGN:
Intervention Model Description: The patients will be divided randomly by a computer-generated randomization table into two equal groups.
Who Masked: Investigator
Masking Description: According to randomization, the anesthesiologist is informed about the ventilation mode but the surgeons are absolutely blind. The surgeons will perform the RIRS without knowing the type of ventilation mode.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Ventilatation Mode (Active Comparator): SV mode is defined according to the mechanical ventilator parameters (patients' age and weight) Standard ventilation mode is defined as 8-10 mL/kg tidal volume and 10-15 respirations/min. No changes were made in the inspiratory expiratory ratio (1:2), FiO2, and positive end-expiratory pressure (PEEP) parameters
  Interventions: Procedure: Changing mechanic ventilatation parameters
- High Ventilatation Mode (Active Comparator): Hv mode is defined as the tidal volume decreased to 6-8 mL/kg and the frequency is increased to 15-18 respirations/min. No changes were made in the inspiratory expiratory ratio (1:2), FiO2, and positive end-expiratory pressure (PEEP) parameters
  Interventions: Procedure: Changing mechanic ventilatation parameters

INTERVENTIONS:
Procedure: Changing mechanic ventilatation parameters — The tidal volume and respiration frequency were determined by the MV according to patient's age and weight with end-tidal CO2 levels of 30-35 mmHg. Standard ventilation mode was defined as 8-10 mL/kg tidal volume and 10-15 respirations/min. During HV mode, the tidal volume was decreased to 6-8 mL/kg and the frequency was increased to 15-18 respirations/min. No changes were made in the inspiratory expiratory ratio (1:2), FiO2, and positive end-expiratory pressure (PEEP) parameters.

SUMMARY:
RIRS (Retrograde Intrarenal Surgery) has been accepted as a first-line treatment option for urinary stones smaller than 2 cm and is generally performed under general anesthesia to manipulate respirator-related renal mobility. Many surgeons prefer general anesthesia during RIRS to minimize respiration-related renal mobility. Standard mechanical ventilation settings were still inadequate to limit renal mobility and the surgeons tried to find the most effective ventilation mode to minimize renal mobility.

DETAILED DESCRIPTION:
A standard general anesthesia protocol is given to all patients by the same anesthesiologist. A Drager Primus (Germany) mechanic ventilator (MV) is preferred for general anesthesia. The MV will determine the tidal volume and respiration frequency according to the patient's age and weight with end-tidal CO2 levels of 30-35 mmHg. Standard ventilation mode is 8-10 mL/kg tidal volume and 10-15 respirations/min. During HV mode, the tidal volume will decrease to 6-8 mL/kg and the frequency will increase to 15-18 respirations/min. No changes are made in the inspiratory expiratory ratio (1:2), FiO2, and positive end-expiratory pressure (PEEP) parameters. The ventilation mode of the mechanic ventilator (SV or HV) is determined via randomization software before the surgery. According to randomization, the anesthesiologist is informed about the ventilation mode but the surgeons are absolutely blind. A high ventilation mode is formed by increasing the respiration frequency and decreasing the study's tidal volume. The aim of the study was to evaluate the effect of this mode on the efficacy and safety of RIRS.

ELIGIBILITY:
Inclusion Criteria:

Patients who underwent RIRS with kidney stones older than18 y.o

Exclusion Criteria:

Patients younger than 18 years old Patients with a known respiratory disease Patients with a renal anomaly Proximal ureteral stones, or stones with multiple locations The patients who underwent previous ipsilateral percutaneous nephrolithotomy and/or open renal surgery were excluded from the study.

Ages: 18 Years to 86 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-02-25 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
perioperatively data of RIRS procedure according to different ventilatation modes | During the surgical procedure
  perioperatively data including e.g. operation time
Complicatation of perioperatively during RIRS | During the surgical procedure
  The presence of perioperative bleeding, perioperative bleeding, ureteral perforation, bladder perforation, ureteral avulsion

SECONDARY OUTCOMES:
Post operative success rates | At the postoperative first month of surgery
  The stone free status and residue stone volume according to CT
Post operative complication | From postoperative first day to postoperative 1. month
  Postoperative complication status including urosepsis, fever, renal colic, flank pain, bleeding and stent migration etc.

CONTACTS AND LOCATIONS:
Overall Officials: Cagri Dogan, Asst.Prof., Study Chair — Namik Kemal University; Cenk Murat Yazici, Prof.Dr., Principal Investigator — Namik Kemal University
Locations (1):
- Cagri Dogan, Tekirdağ, Please Select:, Turkey (Türkiye)

REFERENCES:
- [Derived] Dogan C, Sahin A, Akgul HM, Yazici CM, Keles A, Ates H, Seramet S. Does High Ventilation Mode Affect the Success Rates of Retrograde Intrarenal Surgery? A Single-Blind Randomized, Prospective, Single-Center Study. J Endourol. 2023 Nov;37(11):1169-1173. doi: 10.1089/end.2023.0303. Epub 2023 Sep 25. PMID 37650806